CLINICAL TRIAL: NCT00051857
Title: Virtual Function Anatomy (VFA)
Brief Title: MRI Study of Musculoskeletal Function
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 030060; 03-CC-0060
Record Dates: First submitted 2003-01-16; First posted 2003-01-17 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01-23

CONDITIONS: Abnormalities; Imaging; Patellofemoral Pain Syndrome
Keywords: Patello-Femoral; Knee; Motion; MRI; Kinematics; Natural History
MeSH Terms: conditions — Congenital Abnormalities; Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Healthy Controls: Subjects 5 years old and up with musculoskeletal impairment, pathology, or variant.
- 2/Healthy Volunteers: Subjects 5 years old and up without musculoskeletal impairment, pathology, or variant.

SUMMARY:
This study will use magnetic resonance imaging (MRI) and ultrasound images to study how muscles, tendons, and bones work together to cause motion. The procedure is one of several tools being developed to characterize normal and impaired musculoskeletal function, with the goal of developing improved methods of diagnosis and treatment of movement disorders.

Healthy normal volunteers must be age 5 to unlimited, with or without joint impairment, may be eligible for this study. Volunteers with joint impairment may not have serious injury to the joint being studied, previous surgery on the joint being studied, or extreme pain at the joint being studied.

MRI uses a strong magnet and radio waves to create images of the inside of the body. The subject lies on a long narrow couch inside a metal cylinder (the scanner) for up to 3 hours while the scanner gathers data. Earplugs are worn to muffle loud noises caused by electrical switching of radiofrequency circuits used in the scanning process. A special pad or tube may be placed over or around the region being scanned to improve the quality of the data. The subject will be asked to repeatedly move a specific joint, such as the knee, for brief periods, usually less than 5 minutes. The subject can communicate via intercom with the person performing the study at all times during the procedure, and may request to stop the study at any time.

DETAILED DESCRIPTION:
The overall goal of this technology development initiative is to greatly advance the clinical diagnosis and treatment of musculoskeletal impairments as they relate to joint function. The primary focus of this protocol is to initially develop and ultimately validate a combined set of tools (virtual functional anatomy - VFA) that will enable the accurate and precise measurement, analysis and visualization of three-dimensional (3D) static and dynamic musculoskeletal anatomy (e.g., bone shape, skeletal kinematics, tendon and ligament strain, muscle force, and joint space) from imaging data. We plan to merge and extend our existing MR imaging and analysis capabilities with ultrasound imaging and analysis for the development and implementation of a highly accurate, imaging-based measurement and analysis technique for the non-invasive quantification of complete joint anatomy and tissue dynamics during functional movements. In short, we plan to develop a method for creating 3D digital images of loaded and moving joint tissues (bone, cartilage, muscle, and connective tissues) that reveal joint contact patterns and tissue loads. In conjunction with building this tool, we will evaluate the variability of bone shape across subjects, the sensitivity of defined joint posture (translation and rotation of one bone relative to another) to osteo-based coordinate system definition, and the ability to ultimately use these tools to document and evaluate the function of normal and impaired joint structures (e.g., ACL rupture, patella tracking syndrome...) under simulated conditions experienced during activities of daily living.

The principal investigator has previously developed and tested the primary component in the VFA package, cine-phase contrast and fast-phase contrast (fast-PC) MR imaging, demonstrating both to be highly accurate and precise in the measurement of normal 3D knee joint kinematics and biceps femoris strain. Additional investigators have previously developed techniques for imaging musculoskeletal structures using ultrasonography, demonstrating these techniques to be, likewise, highly accurate and precise in the measurement of biomechanical properties of the soft tissues surrounding the knee and the tendons of the quadriceps femoris. Under this protocol we propose to develop additional numerical reconstruction, image analysis, and display methods and test the applicability of fast-PC MR and ultrasound imaging to the study of various normal and impaired joints (e.g., ankle, wrist, and knee). This development process will require data from human volunteers obtained from both static and dynamic MR and ultrasound images.

This development process will require data from human subjects obtained from both static and dynamic MR and ultrasound images. This development is being guided by our philosophy that impaired joint function likely occurs due to abnormal bone shape, abnormal musculoskeletal movements and forces, or both abnormal bone shape and musculoskeletal movements and forces. Thus, our long-term vision is to non-invasively quantify the in vivo 3D joint kinematics, bone shapes and tissue loads for both the impaired and normal volunteer populations, translate the methods and findings into interventional research and ultimately into common clinical practice.

ELIGIBILITY:
* INCLUSION CRITERIA:

Affected Participants:

* Must be between the ages of 5-95 years.
* Minors < 18 years of age, they must be capable of providing assent (verbal or written) with parental or legal guardian permissions obtained.
* Adults 18 >= years of age, they must be able to provide informed consent.
* Have the presence of a bone, muscle, soft tissue, connective tissue injury, impairment or related muscular skeletal system pathology.
* Ability to have an MRI Scan.

Healthy Volunteer Participants

* Must be between the ages of 5-95 years.
* Minors < 18 years of age, they must be capable of providing assent (verbal or written) with parental or legal guardian permissions obtained.
* Adults 18 >= years of age, they must be able to provide informed consent.
* Ability to have an MRI Scan.

EXCLUSION CRITERIA:

Affected Participants:

-For the MR imaging portion of this study, all participants must complete the NIH Diagnostic Radiology screening questionnaire. If any potential contraindication is found, either the volunteer s doctor (with knowledge of the potential contraindication) or the radiology department at the NIH will be contacted to determine if the potential contraindication would exclude them from the specific MR scans being proposed.

Healthy Volunteer Participants

* Any relevant medical problems
* Clinical signs of an impairment in the joint/limb being studied.
* Any serious injury to the joint/limb being studied, previous surgery on the joint/limb being studied or extreme pain at the joint/limb being studied.
* Neurologic Pathology affecting the muscular skeletal system
* For the MR imaging portion of this study, all participants must complete the NIH Diagnostic Radiology screening questionnaire. If any potential contraindication is found, either the volunteer s doctor (with knowledge of the potential contraindication) or the radiology department at the NIH will be contacted to determine if the potential contraindication would exclude them from the specific MR scans being proposed.

Ages: 5 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be primarily recruited from the greater Washington DC area.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2003-03-05 (Actual)

PRIMARY OUTCOMES:
Dynamic MRI measures of in vivo tissue velocity, bone and muscle, during dynamic tasks of knee flexion/extension | End of study
  MRI techniques to non-invasively measure the 3D in vivo musculoskeletal kinematics, bone shapes, and muscle-tendon lengths in the joints of normal volunteers and healthy volunteers with specific joint impairments.

SECONDARY OUTCOMES:
B-mode ultra-sound of muscles and bones that compose the knee joint | End of study
  Ultrasound techniques to non-invasively measure the 3D in vivo musculoskeletal kinematics, bone shapes, and muscle-tendon lengths in the joints of normal volunteers and healthy volunteers with specific joint impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Frances T Gavelli, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
If other investigators wish to use these data, IRB approval will be sought prior to any data sharing. Data sharing will be done under a waiver of informed consent if (1) the previously signed consent form lacked data sharing information or (2) the consent form contained this information and the participant did not ask that his/her data not be shared. Waiver of consent meets the criteria set out in 45 CFR 46.116(d):@@@@@@@@@@@@The research and data sharing involves no more than minimal risk to the subjects.@@@@@@@@@@@@The waiver or alteration will not adversely affect the rights and welfare of the subjects. Data and samples will have personally identifying information removed.@@@@@@@@@@@@The research could not practicably be carried out without the waiver or alteration.@@@@@@@@@@@@Whenever appropriate, the subjects will be provided with additional pertinent information after participation.
Supporting Information: CSR
Time Frame: Data will be shared through data sharing agreements.@@@@@@@@@@@@The start and end date will be determined by the data sharing agreement.
Access Criteria: Data will be shared stripped of PII and with IRB approval.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-CC-0060.html